

# LETTER OF INFORMATION AND CONSENT TO PARTICIPATE IN A RESEARCH STUDY

TITLE: Evaluating Community Garden Programs as Environmental Health Interventions in Mississauga

## PRINCIPAL INVESTIGATOR:

Vasanti Malik, MSc, ScD Assistant Professor, Department of Nutritional Sciences, Temerty Faculty of Medicine University of Toronto C. David Naylor Building, 2nd Floor, Room 208 6 Queen's Park Cres. Toronto, ON, M5S 3H2 Tel: 416 978-5556

Email: vasanti.malik@utoronto.ca

# **Co-Principal Investigator:**

Britt McKee, MES, OCT Executive Director, Ecosource 2-5070 Fairwind Drive Mississauga, ON L5R 2N4 Tel: 905-274-6222 ext 304

Email: bmckee@ecosoure.ca

## INTRODUCTION

You are invited to be part of a research study. Before you decide to participate, it is important that you read and understand this research consent form. This form contains all the information you need to decide whether you want to participate in the study. If you have any questions, ask the principal investigator or study personnel. The study principal investigator is Dr. Vasanti Malik; you can find her contact information above. You should not sign this form until you are sure you understand the information. Your participation is voluntary. You might also want to discuss this study with your family doctor, a family member or close friend. If you decide to join this study, it is important that you are as accurate as possible about your health history and any medications/products (including natural health products) you are taking. This helps us keep you safe.

You are being asked to participate in a 26-week intervention involving community gardening and cooking classes with nutrition and type 2 diabetes education included. In addition, you are being asked to complete questionnaires (demographic/lifestyle) at baseline (start of the study), 12 weeks (mid-point of the study) and 26 weeks (end of the study). In addition, there will be optional pre- and post-implementation focus groups and post-intervention interviews. All



information will be stored in a secure University of Toronto online storage service. All participants will receive compensation (e.g. gift cards) for their time. All focus groups/interviews will be approximately 60-90 minutes in length and conducted by a research team member in English. Focus groups/interviews will take place either in-person or online at a time that will be convenient for you. Focus groups will be recorded on Zoom if online or using a voice recorder if in person. Voice recordings will be anonymized and stored on a secure University of Toronto online storage service, and transcripts will be analyzed on NVivo which is a qualitative data analysis (QDA) computer software package produced by QSR International.

As part of the 26-week intervention there will be an option to participate in a photovoice project. All participants will receive disposal cameras to document their learning through photography and accompanying image captions. Content analysis of the photographs will be conducted with transcripts of group discussions and image captions analyzed on NVivo. Participants in this part of the study have the option to opt in to a group exhibition of their photographs post-intervention. Please see the supplemental consent form for the photovoice component of the project, if interested in participating. This completed consent form must be signed and provided to the team prior to participation in this study.

## **BACKGROUND**

Peel has one of the highest rates of Type 2 Diabates (T2D) in Ontario. Individuals with T2D have a higher risk of cardiovascular diseases (CVD), kidney disease, lower limb amputation and vision loss compared to the general population. Excess body weight, poor diet, and physical inactivity are key contributors to T2D risk, and are influenced by several factors including structural inequities and our built and food environments. There is an urgent need for local and practical T2D prevention strategies in Peel to ensure the health and quality of life of its residents. A healthy diet and lifestyle are important for precenting chronic diseases, such as T2D.

The Evaluating Community Gardens as Environmental Health Interventions in Mississauga project aims to assess how community gardening can improve health outcomes in Mississauga's priority communities. Building on Ecosource's successful community garden program, the overarching aim of our proposed project is to evaluate community gardening as a potential environmental health intervention for T2D prevention in Mississauga. Existing research suggests that community gardening positively impacts diet quality and physical activity levels, both of which reduce T2D risk. Ecosource's data supports these findings, with participants reporting lower grocery costs, access to culturally relevant foods, and increased outdoor activity, along with other co-benefits such as stronger community ties.

## **OVERALL PROJECT AIMS**

• Aim 1: To deliver a 26-week revised community garden program that integrates education on T2D and cardiometabolic disease prevention.



- Aim 2: To evaluate the impact of the revised program on key T2D risk factors, including
  diet quality and physical activity, and its alignment with Mississauga's Healthy City
  Strategy by improving access to healthy foods and green spaces [1].
- Aim 3: To share the knowledge gained from the evaluation to inform future community gardening initiatives.

## WHAT WILL I NEED TO DO FOR THIS STUDY?

We are inviting you to participate in Aim 1, 2 and 3 for this study. This will involve:

- 1. Participate in a 26-week community gardening and cooking program with nutrition and T2D diabetes education:
  - Weekly sessions will be led by Ecosource and take place in community gardens across different sites in Mississauga and at Ecosource's teaching kitchen located at Hurontario and Eglinton.
  - Diabetes education sessions will take place once per month (6 times/program) and will be led by subject matter experts including dietitians/diabetes educators. The delivery format for these sessions may be virtual or in-person depending on the topic covered and participant availability.
  - Participants will be invited to a WhatsApp Community Chat to stay motivated and engaged with the study over the 26-week period.
- 2. Complete 1 CANRISK questionnaire at baseline and 3 additional questionnaires to assess diet quality, physical activity, and community belonging at baseline, 12 weeks and 26 weeks.
- 3. Participate in an optional photovoice project to document your experience in the intervention by taking photographs during the 26-week program. Participants in this part of the intervention will receive a disposable camera or use of an Ecosource-owned iPad for the purpose of taking photographs. Participants will also be asked permission to use their photographs in dissemination of results including a public exhibition to share study findings. Please see the supplemental consent section following this form if interested in participating in the photovoice project.
- 4. Participate in pre- and/or post-implementation focus groups and interviews (approximately 60-90 minutes) to help develop the program (pre-implementation) determine the effectiveness of the intervention (post-intervention). Participants who participate in a focus group/interview will receive a \$25 gift card.

To express your interest in the <u>optional</u> activities (#3 and #4 above), please indicate by checking the boxes below. Please note by indicating your interest you <u>may</u> be selected for the activity, but participation is not guaranteed.

| YES, I would like to be contacted to participate in a pre-implementation focus group to |
|---|
| help co-create the program. |
| YES, I would like to be contacted to participate in a post-implementation focus group |
| or interview. |



YES, I would like to participate in the photovoice project as part of the 26-week program.

Please see the supplemental consent section following this form.

## PARTICIPANT RECRUITMENT

You have been recruited for this study as you are an adult (18 years of age or over) without chronic conditions that prevent safe participation. Participation in this study will not affect your access to or ability to participate in University of Toronto and Ecosource programs and activities.

## **BENEFITS & RISKS**

The risks involved in this study are minimal. Despite this, there is still a possibility that you may experience different risks as a result of your participation, however, steps will be taken to minimize and manage these risks, as outlined below.

Psychological/emotional risks (e.g., feeling uncomfortable, embarrassed, or upset): There is a possibility of psychological/emotional risks when participants complete the focus group/interview sessions as participants will be asked to share their personal opinions on the different aspects of the study. To minimize this risk, the questions asked during these sessions will not be of a sensitive matter and will be reviewed by a community advisory committee comprising of subject matter experts and Peel community members. Participants may also experience psychological/emotional risks when answering the questionnaires. However, the questionnaires are non-invasive and you will have the option to complete them privately or with the support of trained staff in a private setting. Participants will be provided with resources should they experience any psychological/emotional risks. Such as resources outlined in the Canadian Mental Health Association Peel Dufferin website: https://cmhapeeldufferin.ca/programs-services.

Physical risks (e.g., any bodily contact or administration of any substance): There is a possibility of physical risks when participants engage in gardening and cooking activities. Ecosource has a comprehensive health and safety program for all gardening and cooking activities to minimize physical harm, which includes safety training, weather guidelines, food safety procedures, and staff certifications such as first aid, food handling and vulnerable sector checks. To minimize physical harm while gardening, participants will be instructed to work at their own pace and be provided with gardening gloves/hats and have access to water. In addition, food prepared through the program will follow the dietary recommendations from Canada's Food Guide/Diabetes Canada clinical practice guidelines. While we do not expect adverse side effects from the consumption of food prepared following these guidelines and the advice of dieticians/diabetes educators, we will monitor safety and adverse events during the study.

**Cybersecurity:** Potential breaches to cybersecurity during virtual sessions will be minimized by using a password protected Zoom account and potential breaches to confidentiality regarding health status or personal information will be minimized by a series of steps to maintain data



security (e.g. de-identifying data, using password protected computers, and limiting data access).

## **COMPENSATION**

Participants who take part in this study will be provided with compensation for their time according to the following schedule. Participants will be given a gift card that incrementally increases in value at each stage of the study.

- Upon program start and completion of baseline questionnaires, participants will be given a \$20 gift card.
- Upon completion of 12 weeks of the program and second questionnaire, participants will be given a \$30 gift card.
- Upon completion of 26 weeks of the program and last questionnaire, participants will be given a \$40 gift card.

In addition, participants who participate in a pre- or post-implementation focus group/interview will receive an additional \$25 gift card. Similarly, participants who participate in the photovoice project will receive an additional \$25 gift card.

#### WITHDRAWAL

Participation in this study is voluntary. You may refuse to participate and/or decline to answer any question in any part of the study without negative consequences. If you wish to withdraw your information, this will be done automatically without any questions from the project team. If you choose to withdraw, all of your data collected will be deleted. The project team will not be able to withdraw information from the study one week after it has been collected.

## CONFIDENTIALITY

The questionnaires are being conducted for the purpose of this study and all participants will not be named. All audio recordings will be stored on an encrypted password protected cloud server and deleted from any hard drives and personal cloud storage once transcribed. Digital identifiable focus group/interview transcripts will be stored for 7 years on password protected encrypted University of Toronto servers only accessible to the Principal Investigator. Scanned copies of consent forms will also be retained for 7 years, and hard copies will be destroyed.

## **CONTACT INFORMATION**

If you have any questions about this study, please feel free to contact the Principal Investigator, Vasanti Malik, at vasanti.malik@utoronto.ca or (416) 978-5556.



This study has been reviewed and received ethics approval from the University of Toronto (Human Study REB 00048687). If you have questions regarding your rights as a research participant, contact in the first instance:

Research Oversight and Compliance Office – Human Research Ethics Program 27 King's College Circle Toronto, ON M5S 1A1 at ethics.review@utoronto.ca or 416-946-3273

## **FEEDBACK AND PUBLICATION**

Results of this study may be used in publications and presentations. Your data will be handled as confidentially as possible. If results of this study are published or presented, individual names and other personally identifiable information will not be used. To minimize the risks to confidentiality, your personal information will be kept safe. We may share the data collected from you for use in future research studies or with other researchers – if data collected about you is shared, we will remove any information that could identify you before sharing it.

All participants will be able to view the results. Only aggregate findings and no individual responses will be reported. You can request the executive summary by emailing Vasanti Malik at vasanti.malik@utoronto.ca

# STATEMENT OF CONSENT

I have read and understood the above information. I have received a copy of this form. I agree to participate in this study.

| Name of Participant: | |
|----------------------------------------|---|
| Signature of Participant: | |
| Date: | |
| Name of Person Obtaining Consent: | - |
| Signature of Person Obtaining Consent: | |
| Date: | |

# SUPPLEMENTAL LETTER OF INFORMATION AND CONSENT FOR PHOTOVOICE PROJECT



Please only complete this section if you indicated you would like to participate in the optional photovoice project as part of the 26-week intervention.

## **INTRODUCTION**

Photovoice is a participatory research method that combines photography and social action. It gives people a voice by letting them document their experiences and share their perspectives through photos. It's often used in community-based research, public health, education, and social work to empower individuals, raise awareness, and influence policy.

You will be asked to take photographs during participation in weekly gardening and cooking activities to document your learning and experience. In addition, you will be asked to describe the photographs you take in your own words. Group discussions will be held at 12 weeks and 26 weeks to explore the meaning of the photographs. These discussions will be recorded and transcribed with transcripts analyzed on NVivo which is a qualitative data analysis (QDA) computer software package produced by QSR International. All participants will receive disposable cameras or Ecosource-owned iPads to take photographs for the project.

## PARTICIPANT RECRUITMENT

You have been recruited for this study as you are an adult (18 years of age or over) without chronic conditions that prevent safe participation.

#### WHAT WILL I NEED TO DO FOR THIS PHOTOVOICE PROJECT?

We invite you to take part in a photography activity as part of the 26-week community gardening and cooking program described in the previous consent form. This activity includes:

- Attending a training session on how to take photographs and follow the project's ethical guidelines (e.g., getting informed consent from anyone you photograph, not taking photographs of minors, etc.).
- Taking photographs during the program that reflect your experiences, based on the training and ethical guidelines, and writing short captions to explain what the photos mean to you.
- Choosing which photographs, if any, you feel comfortable sharing during group discussions held at weeks 12 and 26 of the program.
- Choosing which photographs, if any, you feel comfortable allowing the project to use in materials such as reports, leaflets, books, postcards (both printed and digital), websites, social media, apps, public exhibitions, and other project-related promotions, including potential media coverage

## **BENEFITS & RISKS**

Photovoice presents specific ethical risks, particularly concerning photo ownership, informed consent, and the protection of confidentiality. These risks include the potential identification of individuals in photographs, unauthorized use or sharing of images, and the inadvertent disclosure of sensitive or private information.



To mitigate these risks, all participants will receive comprehensive training on ethical photography practices, including the importance of obtaining informed media consent and respecting the privacy of others. Participants will be explicitly instructed not to photograph individuals under the age of 18 or any individuals unable to provide informed consent. Written, informed consent will be obtained from every individual who appears in a photograph. Additionally, photographers will be required to sign a release form granting permission for their images to be used in the dissemination of research findings, including public exhibits, academic publications (both print and digital), and presentations.

To further protect participants' identities and confidentiality, all photographs and accompanying narratives will be anonymized. This includes the use of pseudonyms and the exclusion or alteration of any identifying details in captions or narratives. These measures will ensure the ethical handling of visual data and uphold the dignity, autonomy, and privacy of all individuals involved.

#### **COMPENSATION**

Participants who take part in the photovoice project will be provided with compensation for their time. A \$25 gift card will be available to you if you submit a minimum of one eligible photo and caption to the project **and** attend one group discussion of the photographs.

# WHAT AM I AGREEING TO

As part of this project, you will produce photographs and text. As the creator of the photographs and text, you own them and keep the copyright to them. This form gives the partners involved in the project permission (which is called a licence) to keep and use copies of the images and text for the purposes of the project. You will be able to select which of your photographs and text to give permission to use. If you have chosen photographs and/or captions which describe or refer to things such as your religious or philosophical beliefs, your racial or ethnic origin, your health circumstances, or other such personal information, you understand that this information is considered 'sensitive' and that it is your choice to share.

## HOW I WILL BE CREDITED FOR MY WORK

You will always be credited for your photographs and text, however to protect your confidentiality Ecosource will not use your full name in credit lines. While this consent form will contain your full name, this will never be shared with others outside the project partners stated above. You can choose to be credited for your work with either: your first name, or a pseudonym/alias/nickname you have chosen. This information will be collected on a separate photo release form.

## HOW MY PHOTOGRAPHS WILL BE USED

By agreeing below, you give permission for the project team and its partners to keep and share your photos and captions. These may be used in:



- Project materials like reports, leaflets, books, or postcards (both printed and digital)
- Websites, social media, and apps that are publicly available online
- Public exhibitions
- Promotional materials about the project, including possible coverage by news outlets

You are always in control of what you choose to share. If there's any photo or story you don't want to be used, you are under no pressure to include it. In addition, you can still take part in the project activities even if you choose not to share any of your photos or stories.

#### **ADDITIONAL CONSIDERATIONS**

#### 1. Public Use and Access

If you consent to your photographs and captions being shared publicly, you understand that the project team cannot control who views, downloads, or uses the content once it has been made available in the public domain.

# 2. Editing and Formatting

The project team may crop, resize, or combine your photographs with text or graphic elements to meet the formatting requirements of various platforms (e.g., print publications, websites, exhibitions). Any such modifications will be made solely for presentation purposes and will not alter the intended meaning of your contribution.

# 3. Right to Withdraw Consent

You retain the right to withdraw your permission to use your photographs and captions at any time by notifying the principal investigator in writing.

- o Upon withdrawal, the project team will cease any further use of your materials.
- Please note that withdrawal cannot apply retroactively to content already shared, published, or archived in public domains.

## 4. Limitations on Withdrawal

While the project team will discontinue future use of your contributions upon withdrawal, it may not be possible to remove materials already published or distributed. However, your photographs and captions will not be used in any future publications or reprints following the withdrawal of consent.

# 5. Retention of Copyright

You will retain full ownership and copyright of your photographs and captions. You are free to use your content independently and without restriction.

## 6. Limitations on Control Over Public Use

Although the project team will adhere to the agreed-upon terms of use, once your content is made publicly accessible, it may be copied, shared, or used by others without the knowledge or permission of the project team. The team cannot be held responsible for any such third-party use.

# 7. Data Storage and Privacy

Your photographs, captions, and any associated personal information will be stored securely by the project team in accordance with applicable data protection and privacy regulations.



# 8. Third-Party Sharing

Your contributions may be shared with partner organizations or collaborators, but only for the purposes outlined in the research study and in line with the consent you have provided.

## CONFIDENTIALITY

The photographs and captions collected as part of this project will be attributed to first names or pseudonyms only to protect the confidentiality of participants. Audio recordings of group discussions will be stored on an encrypted password protected cloud server and deleted from any hard drives and personal cloud storage once transcribed. Discussion transcripts will be stored for 7 years on password protected encrypted University of Toronto servers only accessible to the Principal Investigator. Scanned copies of consent forms will also be retained for 7 years, and hard copies will be destroyed.

## **CONTACT INFORMATION**

If you have any questions about this project, please feel free to contact the Principal Investigator, Vasanti Malik, at vasanti.malik@utoronto.ca or (416) 978-5556.

This study has been reviewed and received ethics approval from the University of Toronto (Human Study REB 48687). If you have questions regarding your rights as a participant, contact in the first instance:

Research Oversight and Compliance Office – Human Research Ethics Program 27 King's College Circle Toronto, ON M5S 1A1 at <a href="mailto:ethics.review@utoronto.ca">ethics.review@utoronto.ca</a> or 416-946-3273

## **FEEDBACK AND PUBLICATION**

Results of this project, including your photographs, may be used in publications and presentations. Your data will be handled as confidentially as possible. If results of this study are published or presented, individual names and other personally identifiable information will not be used, except where consented to above. To minimize the risks to confidentiality, your personal information will be kept safe. We may share the data collected from you for use in future research studies or with other researchers – if data collected about you is shared, we will remove any information that could identify you before sharing it.

All participants will be able to view the results. Only aggregate findings and no individual responses will be reported. You can request the executive summary by emailing Vasanti Malik at <a href="mailto:vasanti.malik@utoronto.ca">vasanti.malik@utoronto.ca</a>

# STATEMENT OF CONSENT



I have read and understood the above information. I have received a copy of this form. I agree to participate in this the photovoice component of the study.

| Name of Participant: |
|----------------------------------------|
| Signature of Participant: |
| Date: |
| Name of Person Obtaining Consent: |
| Signature of Person Obtaining Consent: |
| Date: |